CLINICAL TRIAL: NCT06409494
Title: A PhaseⅠ, Randomized, Observer-blinded, Active Comparator, First-in-human Clinical Trial to Evaluate Safety and Tolerability of Herpes Zoster Vaccine EuHZV in Healthy Adults Aged 50 to 69 Years
Brief Title: Clinical Trial to Evaluate EuHZV in Healthy Adults Aged 50 to 69 Years
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EuHZV_101
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Varicella Zoster Virus Infection; Herpes Zoster
Keywords: EuHZV; HZV; Varicella Zoster Virus; Herpes Zoster
MeSH Terms: conditions — Varicella Zoster Virus Infection; Herpes Zoster; Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HZV-1 (Experimental): Biological: EuHZV Healthy adults received 0.5mL single intramuscular dose on Visit 2(Day 0) and Visit 4(day 56).
  Interventions: Biological: EuHZV
- HZV-2 (Experimental): Biological: EuHZV Healthy adults received 0.5mL single intramuscular dose on Visit 2(Day 0) and Visit 4(day 56).
  Interventions: Biological: EuHZV
- Shingrix (Active Comparator): Biological: Shingrix Healthy adults received 0.5mL single intramuscular dose on Visit 2(Day 0) and Visit 4(day 56).
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: EuHZV — Drug(injection)
  Arms: HZV-1; HZV-2
Biological: Shingrix — Drug(injection)
  Arms: Shingrix

SUMMARY:
Phase 1 clinical trial to evaluate the safety of HZV-1 and HZV-2 vaccines in healthy adults aged 50 to 69 years who have voluntarily given written consent to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult men and women between the ages of 50 and 69 years old
2. Have a body mass index (BMI) of at least 18 kg/m2 and no more than 30 kg/m2 at the screening visit
3. Men and women who agree to use a highly effective method of contraception (*See section 8.7 of the protocol) (however, not women of childbearing age or men who do not have a spouse (partner) may be enrolled regardless of method of contraception).

   * Women of childbearing potential: Practiced a highly effective method of birth control for 4 weeks prior to the first dose of study medication and agreed to continue to use a highly effective method of birth control for the duration of the study (up to 3 months after the last dose of study medication).
   * Men who have a spouse (partner): Has agreed to use a highly effective method of birth control for the duration of the study (up to 3 months after the last dose of study medication).
4. Agree to refrain from donating blood and transfusions (whole blood, plasma components, platelet components, platelet-plasma components) for the duration of the study.
5. After receiving and understanding a detailed explanation of this clinical trial, voluntarily decide to participate and give written consent.
6. For women of childbearing potential, a negative pregnancy test prior to receiving the investigational drug.

Exclusion Criteria:

1. Clinically significant abnormalities on clinical laboratory tests, electrocardiogram (ECG), or chest x-ray at screening.
2. Positive hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) test results at screening.
3. Active pulmonary infection within 14 days prior to the first dose of investigational medicinal product, or any other significant infectious disease that, in the opinion of the investigator, would render the subject ineligible for participation in the study.
4. Have had an acute febrile illness of 38 degrees or greater within 3 days prior to the first dose of investigational drug
5. Have any of the following conditions, or any serious medical or neuropsychiatric condition that, in the opinion of the investigator, would make them ineligible to participate in this study.

   * Respiratory disease: asthma, chronic obstructive pulmonary disease (COPD), active tuberculosis, or latent tuberculosis.

     * Serious cardiovascular disease: Congestive heart failure, coronary artery disease, myocardial infarction, uncontrolled hypertension, myocarditis, pericarditis, etc.

       * Nervous system disease: epilepsy, seizures (within 3 years prior to first dose of investigational drug), migraine, stroke, cerebral lesions, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, dementia, etc.

         ④ History of malignancy within 5 years prior to the first dose of investigational drug and a history of malignant disease with a high risk of recurrence (skin basal cell carcinoma and squamous cell carcinoma with a minimal risk of recurrence based on clinical judgment may be eligible).

         ⑤ Autoimmune diseases including autoimmune hypothyroidism and psoriasis

         ⑥ Immunodeficiency diseases

         ⑦ Thrombosis at uncommon sites, such as cerebral venous sinus thrombosis and visceral venous thrombosis, and heparin-induced thrombocytopenia or antiphospholipid syndrome

         ⑧ Capillary leak syndrome

         ⑨ Other hepatobiliary, renal, endocrine, urinary, or musculoskeletal diseases deemed clinically significant by the investigator
6. History of allergic reactions or hypersensitivity to any of the components of the investigational drug.
7. History of serious adverse events, serious allergic reactions, or serious hypersensitivity reactions related to vaccination.
8. History of platelet-related or hemorrhagic disease (such as major venous and/or arterial thrombosis with thrombocytopenia), or history of excessive bleeding or bruising after intramuscular injection or venipuncture, or receiving anticoagulant therapy (except that patients may participate if they are using low-dose anticoagulants (e.g., aspirin <100 mg/day) as determined by the investigator).
9. History of systemic urticaria within 5 years prior to the first dose of investigational drug.
10. Have a history of hereditary or idiopathic angioneurotic edema
11. History of organ or bone marrow transplantation
12. History of dependent use of antipsychotics or narcotic analgesics within 6 months prior to the first dose of study medication, or psychiatric or social conditions that, in the opinion of the investigator, would make it difficult to comply with the procedures of this study.
13. Suspected history of drug abuse or alcohol abuse
14. History of varicella or varicella-zoster virus (VZV) vaccination or participation in a varicella or zoster vaccine clinical trial
15. Active antiviral therapy for varicella-zoster virus (VZV) within 1 week prior to the first dose of investigational medication. (e.g., Acyclovir, Valacyclovir, Famciclovir, Ganciclovir, etc.) (however, topical use is allowed)
16. Treatment with immunosuppressive or immunomodulatory agents or chronic steroid use within 6 months prior to the first dose of investigational product.

    ① Immunosuppressants or immunomodulators: Azathioprine, Cyclosporine, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus, Cyclophosphamide, 6-Mercaptopurine, Methotrexate, Rapamycin, Leflunomide, etc.

    ② Systemic steroids: Prednisolone at a dose of ≥10 mg/day for more than 14 consecutive days (topical, inhaled, nasal corticosteroids and eye drops are allowed at any dose).
17. Received any other investigational drug or received an investigational medical device within 6 months of the screening visit.
18. A history of herpes zoster and/or varicella within 10 years of the screening visit, or planned treatment for these conditions during the study period.
19. Have received or plan to receive any other vaccine within 4 weeks prior to or after each dose of investigational product.

    (Allow influenza vaccines and COVID-19 vaccines, but not vaccinations within 14 days before or after receiving an investigational drug)
20. Treatment with immunoglobulins or blood-derived products within 3 months prior to the first dose of investigational medicinal product or planned treatment during the study period
21. Pregnant or lactating women
22. For any other reason deemed by the investigator to be unsuitable as a patient in this study

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of immediate adverse events | within 30 minutes post vaccination
  local and systemic AEs
Occurrence of solicited adverse events | within 7 days post vaccination
  local and systemic AEs
Occurrence of unsolicited adverse events | within 52 weeks post vaccination
  local and systemic AEs
Occurrence of serious adverse events | within 52 weeks post vaccination
  local and systemic AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Eunpyeong St.Mary's Hospital, Seoul, South Korea